CLINICAL TRIAL: NCT03302208
Title: Role of Preoperative Oral Pregabalin in Reducing Inhalational Anesthetic Requirements in Elective Abdominal Hysterectomy Under General Anesthesia: A Randomized Controlled Trial
Brief Title: Preoperative Oral Pregabalin Effect on Inhalational Anesthetic Requirements ln Hysterectomy Under General Anesthesia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nesrine El-Refai (Other)
Responsible Party: Sponsor-Investigator, Nesrine El-Refai, professor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: UTF-9
Record Dates: First submitted 2017-06-29; First posted 2017-10-05 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Hysterectomy
Keywords: General Anesthesia
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pregabalin group (Active Comparator)
  Interventions: Drug: Pregabalin
- placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — Pregabalin capsule 150 mg oral
  Other Names: laryca
  Arms: pregabalin group
Drug: Placebo — Placebo
  Arms: placebo group

SUMMARY:
In this study the investigators hypothesized that preoperative pregabalin tablet (150 mg orally ) may be effective in reducing intraoperative isoflurane requirements needed to maintain intraoperative hemodynamics within ± 20% of baseline measurement and/or attenuates hemodynamic response to endotracheal intubation in female patients ASA I or II , aged 18-60 years, schedule for elective abdominal hysterectomy surgery under general anesthesia.

DETAILED DESCRIPTION:
In this study the investigators hypothesized that preoperative pregabalin tablet (150 mg orally ) would be effective in reducing intraoperative isoflurane requirement needed to maintain intraoperative hemodynamics within ± 20% of baseline measurement and/or attenuates hemodynamic response to endotracheal intubation in female patients ASA I or II schedule for elective abdominal hysterectomy surgery under general anaesthesia.

The investigators aim to compare the efficacy of preoperative oral pregabalin versus placebo in reducing intraoperative isoflurane requirements needed to maintain intraoperative hemodynamic stability (Blood pressure and heart rate within ± 20% of baseline measurements) in female patients ASA I/II undergoing elective abdominal hysterectomy surgery under general anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Female patients, aged 18-60 year scheduled for elective abdominal hysterectomy surgery under general anaesthesia.
* American Society of Anaesthesiology (ASA) physical status I or II.

Exclusion Criteria:

* American Society of Anaesthesiology (ASA) physical status ≥ III.
* Allergy or hypersensitivity to pregabalin.
* Patient on calcium channel blocker or anticonvulsant.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-20 (Actual)

PRIMARY OUTCOMES:
Inhalational anaesthetic drug requirements | an average of 3 hours after induction
  Inhalational anaesthetic requirements to maintain hemodynamic stability (± 20% of the baseline) using MAQUET Flow-I anesthetic machine.

SECONDARY OUTCOMES:
pressor response attenuation | an average of 10 minutes after induction
  Degree of pressor response attenuation
First time for analgesics requirement | postoperative (maximum 6 hours after the end of operation)
  First time for analgesics requirement.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Zamalek, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-31): https://cdn.clinicaltrials.gov/large-docs/08/NCT03302208/Prot_SAP_002.pdf